CLINICAL TRIAL: NCT00660634
Title: The Effect of Angioplasty in Peripheral Arterial Disease on Endothelial Function
Brief Title: Angioplasty in Peripheral Arterial Disease and Endothelial Function
Acronym: PTA-PAD-FMD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss Heart Foundation (Other)
Responsible Party: Dr. med. Marc Husmann/Prof. I Baumgartner, Angiology Div. University Hospital of Berne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 85/2004; SHF2006
Record Dates: First submitted 2008-04-10; First posted 2008-04-17 (Estimated); Last update posted 2008-04-28 (Estimated); Status verified 2008-04

CONDITIONS: Peripheral Arterial Obstructive Disease; Intermittent Claudication
Keywords: Peripheral arterial obstructive disease; Intermittent Claudication; Endovascular treatment; Flow-mediated dilation
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (No Intervention)
- A (Experimental): Endovascular angioplasty/stenting
  Interventions: Procedure: Endovascular Revascularization

INTERVENTIONS:
Procedure: Endovascular Revascularization — Angioplasty/Stenting of femoro-popliteal lesions
  Arms: A

SUMMARY:
To investigate whether endovascular revascualrization of infrainguinal arterial obstructive disease has an effect on brachial artery reactivity

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is a common manifestation of atherosclerosis affecting a large proportion of the aged population. It is associated with a more or less severe impairment in functional activity and with an increased risk of future cardiovascular events. In PAD patients, an increased inflammatory status and a depressed endothelial function, assessed as flow-mediated dilation of the brachial artery have been demonstrated. Moreover, a prognostic value has been found in PAD patients for both inflammatory parameter and flow-mediated dilation (FMD). One of the reasons of the increased inflammatory activation and endothelial dysfunction in PAD patients could be the ischemia-reperfusion injury associated with intermittent claudication. The hypothesis is that repeated episodes of acute inflammation and endothelial dysfunction following ischemia-reperfusion injury linked to intermittent claudication could be in part responsible for the increased inflammatory status and chronically depressed endothelial dysfunction of these patients. Taking into account these considerations, it is reasonable to assume that the correction of leg ischemia by interventional procedure, such as peripheral transluminal angioplasty (PTA) should determine a reduction in inflammatory mediators and an improvement in endothelial function.

The study is a prospective, open, randomised, controlled, single-centre, follow-up evaluation, assessing the efficacy of peripheral catheter interventions in patients with symptomatic PAD on endothelial dysfunction and plasmatic procoagulant activity. Patients will be randomly assigned to immediate revascularization or to no treatment for one month. The assessment of parameters (brachial artery flow-mediated and nitrate-mediated dilation, plasma levels of C reactive protein, fibrinogen, microparticles and coagulation factors) will be performed at baseline and after 4 weeks in both, patients undergoing interventional procedures and in those, who will not be treated.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral arterial disease
* femoro-popliteal lesion
* successful endovascular treatment of lesion

Exclusion Criteria:

* persistent claudication after revascularization in arm A
* inflammatory or neoplastic disease
* pregnancy

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2004-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Improvement of Flow-mediated Dilation | 4 weeks

SECONDARY OUTCOMES:
Improvement of white blood cell count | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Husmann, MD, Principal Investigator — Angiology Division, University Hospital of Berne, Switzerland